CLINICAL TRIAL: NCT00476489
Title: Low Dose (1mcg) ACTH Stimulation Test for Assessment of the Hypothalamo-Pituitary- Adrenal Axis in Patients Treated With Topical Corticosteroids
Brief Title: Does Topical Steroid Treatment Impair the Adrenal Function?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Other Study IDs: 02307EMC
Record Dates: First submitted 2007-05-21; First posted 2007-05-22 (Estimated); Last update posted 2007-05-22 (Estimated); Status verified 2007-05

CONDITIONS: Hypothalamus-Pituitary-Adrenal Axis Assessement; Topical Steroid Therapy in Chronic Skin Diseases
Keywords: secondary adrenal insuffiency; hypothalamus-pituitary-adrenal axis impairement; topical steroids

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine if topical steroids treatment for different skin diseases suppress the adrenal cortisol production.

DETAILED DESCRIPTION:
Adrenocortical suppression is a potential complication of systemic corticosteroid treatement but also of non systemic therapy like topical therapy.

The normalcy of hypothalamic-pituitary-adrenal axis ( HPA axis) of patients with chronic skin diseases like atopic dermatitis, pemphigus or psoriasis which are treated with topical steroids, will be assessed with the low dose (1mcg) adrenocortocotropin ( ACTH) stimulation test. During this test serum cortisol levels are measured before, 30 and 60 mn after intravenous administration of 1mcg of ACTH (synacthen).The results will be compared with age and sex matched subjects with normal HPA axis as assessed by low dose ACTH stimulation test.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving daily topical steroids for at least two weeks on 10% or more of body surface.

Exclusion Criteria:

* patients treated with any form of corticosteroids except topical steroids.
* patients with known pituitary disease
* pregnant patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-05

CONTACTS AND LOCATIONS:
Overall Officials: Avraham Ishay, MD, Principal Investigator — haemek medical center
Locations (1):
- Haemek Medical Center, Afula, Israel